CLINICAL TRIAL: NCT04409249
Title: Prognostic Factors in Pregnant Women With COVID-19
Brief Title: Prognosis in Pregnant With COVID-19
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Aldikactioglu Talmac, MD, Specialist of Obstetrics and Gynecology, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Mtalmacprognosis
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Prognostic Factors; Pregnancy
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Imaging; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: imaging, blood tests — PCR and CT results, hemogram, urea, creatinine, AST, ALT, LDH, D-Dimer, ferritin, lipase, amylase, CRP, procalcitonin, albumin, total protein, coagulation tests-PT, APTT, Fibrinogen-, Troponin T, CK , electrolytes, blood gas, bilirubins

SUMMARY:
COVID-19 is a disease whose development, prognosis mechanism and immune status are still unknown. The aim of the study is to determine the relationship between clinical and laboratory data and the severity of the disease by evaluating the hematological and radiological features of the patients. The secondary aim is to determine the predictive values of clinical and laboratory data for the severity of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant with a diagnosis of COVID-19 between the ages of 18-45

Exclusion Criteria:

* Suspected COVID-19 diagnosis

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Tertiary center data
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
the factors affecting prognosis in pregnant women diagnosed with COVID-19 | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Halkali, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol